CLINICAL TRIAL: NCT01179503
Title: Vitamin D Supplementation, Skeletal Muscle Gene Expression, and Physical Performance in Older Adults
Brief Title: Vitamin D Supplementation and Physical Function in Older Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00011371; R01AG029364-03S1 (NIH)
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Physical Function; Vitamin D Insufficiency
Keywords: vitamin D; physical performance
MeSH Terms: interventions — Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Calcium only (Active Comparator): 1200 mg Calcium per day
  Interventions: Dietary Supplement: calcium
- Vitamin D plus calcium (Experimental): 2000 IU vitamin D plus 1200 mg calcium per day
  Interventions: Dietary Supplement: Vitamin D plus calcium

INTERVENTIONS:
Dietary Supplement: calcium — 600 mg calcium carbonate twice daily (total of 1200 mg/day) for 4 months
  Arms: Calcium only
Dietary Supplement: Vitamin D plus calcium — 1000 IU of vitamin D3 twice daily (for a total of 2000 IU/day) plus 600 mg calcium carbonate twice daily (for a total of 1200 mg/day)
  Arms: Vitamin D plus calcium

SUMMARY:
A growing body of evidence suggests that vitamin D status is important in biologic processes involved in the maintenance of physical function. To advance the investigators understanding of the role of vitamin D in physical function, the investigators will conduct a feasibility pilot study to collect key information to help design a full-scale randomized trial to determine whether vitamin D supplementation will delay declines in physical function. The primary goals of the pilot study are to determine cost-effective strategies for identifying persons at high risk for functional decline with insufficient vitamin D levels, determine the serum vitamin D response to a vitamin D supplementation regimen designed to attain sufficient vitamin D levels, and provide preliminary data of key functional measures (balance, physical performance and muscle power) for the future larger study design. A secondary goal is to begin to examine potential mechanisms by which vitamin D supplementation may enhance physical performance by exploring the effects of vitamin D supplementation on changes in skeletal muscle gene expression.

DETAILED DESCRIPTION:
A growing body of evidence suggests that vitamin D status is important in biologic processes involved in the maintenance of physical function. However, whether remediation of vitamin D insufficiency will improve physical function and the potential mechanisms involved are unclear. Previous vitamin D supplementation trials have produced mixed results with respect to physical function; however, most trials did not specifically recruit individuals who were vitamin D insufficient nor is the potential mechanism of action understood well enough to appropriately select those individuals most likely to benefit. To advance our understanding of the role of vitamin D in physical function, the investigators will conduct a feasibility pilot study to collect key information to help design a full-scale randomized trial to determine whether vitamin D supplementation will delay declines in physical function. The primary goals of the pilot study are to determine cost-effective strategies for identifying persons at high risk for functional decline with insufficient vitamin D levels, determine the serum vitamin D response to a vitamin D supplementation regimen designed to attain sufficient vitamin D levels, and provide preliminary data of key functional measures (balance, short physical performance battery (SBBP) and muscle power) for the future larger study design. A secondary goal is to begin to examine potential mechanisms by which vitamin D supplementation may enhance physical performance and muscle contractility by exploring the effects of vitamin D supplementation on changes in skeletal muscle gene expression using microarrays.

ELIGIBILITY:
Inclusion Criteria:

* Short Physical Performance Battery (SPPB) score of ≥ 4 to < 10
* Vitamin D insufficient (serum 25(OH)D ≥ 10 to < 25 ng/mL)

Exclusion Criteria:

* Serious or uncontrolled chronic disease including: insulin-dependent or uncontrolled diabetes; cancer requiring treatment in past year, except non-melanoma skin cancers; past or current ischemic heart disease, uncontrolled angina, heart failure, peripheral artery disease (PAD), or stroke; chronic respiratory disease; uncontrolled endocrine/metabolic disease; neurological or hematological disease; liver or renal dysfunction; and severe musculoskeletal impairment
* Impaired cognitive function (MMSE ≤ 24)
* Dependent on a cane or walker
* Use of anti-coagulants
* Unwillingness to undergo a muscle biopsy
* Taking prescription vitamin D2 or OCT vitamin D3 supplements of > 1000 IU/d
* Inability or contraindications to consume daily vitamin D and calcium supplements
* Weight loss of ≥ 5% or more in the past 6 months
* Involved in any other intervention

Ages: 70 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in Physical performance | 4 months
  Change in the expanded Short Physical Performance Battery (SPPB) score (composite score including the following: timed 4m walk; time to stand from a chair 5 times without the use of arms; and time to hold side-by-side, semi-tandem, tandem, and one legged stands for the testing of balance)

SECONDARY OUTCOMES:
Skeletal muscle gene expression | 4 months
  Muscle will be obtained from the vastus lateralis using the percutaneous needle biopsy technique. Five µg of RNA will be supplied for each experimental condition to be analyzed. The WFUHS MicroArray Core Facility further purifies the provided RNA over an RNAeasy column and performs all subsequent steps of the GeneChip protocol (cDNA generation, generation of biotinylated cRNA, chip hybridization, and generation of .CEL files).
Change in expanded SPPB balance task time | 4 months
  Change in expanded SPPB balance task time (time to hold side-by-side, semi-tandem, tandem, and one legged stands; max of 30 sec)
Change in narrow 4m walk test of balance time | 4 months
  Change in time to complete narrow 4m walk test of balance (usual pace over 4m while staying between lines of colored tape placed 20cm apart)
Change in 400m walk test time | 4 months
  Change in 400m walk test time (usual pace)
Change in knee extensor power | 4 months
  Change in knee extensor power measured by the Nottingham Power Rig

CONTACTS AND LOCATIONS:
Overall Officials: Denise K Houston, PhD, Study Director — Wake Forest University; Stephen B Kritchevsky, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States